CLINICAL TRIAL: NCT06571396
Title: Perioperative Risk Factors and Nomograms for Participants With Hepatocellular Carcinoma Receiving Neoadjuvant Immunotherapy or Conversion Therapy
Brief Title: Perioperative Risk of Immunotherapy Based Neoadjuvant and Conversion Therapy for Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-2024(ZM)-1324
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Hepatocellular; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Feces, blood, urine, tissue, pathological sections

SUMMARY:
This study aims to retrospectively collect a cohort of participants with hepatocellular carcinoma who received immunotherapy-based neoadjuvant/translational treatment. A multi-dimensional and multi-method analysis plan will be adopted. The goal is to provide solutions for better application of neoadjuvant immunotherapy and to offer better evidence for conducting prospective clinical research on hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is indeed a significant health concern, especially in regions like China where its incidence and mortality rates are notably high. Radical resection is the main method for curing HCC. However, about 64% of HCC participants are diagnosed at mid to late stages, making surgical resection unsuitable as the first choice. Additionally, the short-term recurrence rate after HCC surgery is relatively high, with a five-year recurrence and metastasis rate reaching 70%. Therefore, increasing the radical resection rate and reducing the postoperative recurrence rate are key measures to improve prognosis.

With the development of tumor genomics and immunology, systematic treatment based on immune checkpoint inhibitors (ICIs) has shown remarkable efficacy in improving HCC prognosis. The application of ICIs in perioperative treatment of solid tumors can effectively reduce tumor burden while expanding the immune effect of tumor antigens, thereby increasing resection rates and reducing recurrence rates.

Currently, neoadjuvant immunotherapy has achieved good treatment outcomes in lung cancer, esophageal cancer, and gastric cancer. However, the increased antitumor treatment may lead to potential treatment side effects. For neoadjuvant immunotherapy in solid tumors, preoperative treatment can pose perioperative risks such as tissue edema, adhesions, and excessive bleeding during surgery. Due to the hidden effects of some immune therapy adverse reactions, these perioperative risks require particular attention and research.

Neoadjuvant immunotherapy for HCC is still in its infancy, with a limited number of cases reported by various centers, and there are currently no large-sample clinical studies available.

The investigators intend to establish a cohort of HCC participants undergoing neoadjuvant/conversion treatment. It will employ a multidimensional and multi-method analysis plan to systematically investigate the perioperative risks associated with immunotherapy in these participants, aiming to provide solutions for better application of neoadjuvant immunotherapy in HCC, while also offering improved evidence for the conduct of prospective clinical research in HCC.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following conditions in order to be enrolled in this study:

1. Voluntarily participate in this study and sign an informed consent form.
2. Participants diagnosed with HCC through pathological histology/cytology or clinically diagnosed with HCC according to the Diagnosis and Treatment Guidelines for Primary Liver Cancer (2024 Edition).
3. Received immunotherapy based neoadjuvant or conversion therapy.
4. Complete recovery from surgical resection within 4 weeks prior to enrollment.
5. Child Pugh liver function rating A or B (≤ 7 points).
6. ECOG PS score was 0-1 points.
7. Expected survival time ≥ 12 weeks.
8. If suffering from hepatitis B virus (HBV) infection, it is necessary to be willing to receive antiviral treatment throughout the study period (according to the diagnostic and treatment guidelines, such as entecavir) and regularly monitor it; Hepatitis C virus (HCV) ribonucleic acid (RNA) positive subjects must receive antiviral treatment according to the diagnosis and treatment guidelines, and their liver function must be within CTCAE1 level elevation.

Exclusion Criteria:

If a subject meets any of the following conditions, they will not be allowed to enter this study:

1. Known hepatobiliary carcinoma, sarcoma like hepatocellular carcinoma, combined hepatocellular-cholangiocarcinoma and fibrous layer cell carcinoma; Within 5 years or simultaneously suffering from other active malignant tumors other than hepatocellular carcinoma (excluding cured skin basal cell carcinoma and cervical carcinoma in situ).
2. There are uncontrollable extrahepatic metastases, such as lung and brain metastases (EHS).
3. Participants who are preparing to undergo or have previously received organ or allogeneic bone marrow transplantation.
4. Participants who are currently accompanied by interstitial pneumonia or interstitial lung disease, or have a history of interstitial pneumonia or interstitial lung disease that requires hormone therapy in the past, other pulmonary fibrosis, organized pneumonia (such as bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or subjects with evidence of active pneumonia or severe lung function impairment seen on chest computed tomography (CT) images during screening, are allowed to have radiation induced pneumonia in the radiation field; Active tuberculosis
5. Currently, there is active autoimmune disease or a history of autoimmune disease that may recur (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects that can be controlled only through hormone replacement therapy can be included]); Subjects with skin diseases that do not need systematic treatment, such as vitiligo, psoriasis, alopecia, controlled type I diabetes that receive insulin treatment, or childhood asthma that has completely alleviated without any intervention after adulthood can be included; Asthma subjects who require medical intervention with bronchodilators cannot be included.
6. Suffering from hypertension and unable to achieve good control through antihypertensive drug treatment (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg) (based on the average BP reading obtained from ≥ 2 measurements), it is allowed to achieve the above parameters through the use of antihypertensive therapy; Previously experienced hypertensive crisis or hypertensive encephalopathy.
7. Participants with moderate to severe ascites with clinical symptoms who require therapeutic puncture or drainage, or whose Child Pugh score is greater than 7 (excluding those who only show a small amount of ascites on imaging but do not have clinical symptoms); Uncontrolled or moderate to equal amounts of pleural effusion and pericardial effusion.
8. There are clinical symptoms or diseases of the heart that cannot be well controlled, such as: (1) According to the standards of the New York Heart Association (NYHA), level II or above cardiac insufficiency or cardiac ultrasound examination: LVEF (left ventricular ejection fraction)<50%; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year prior to the start of the research treatment; (4) Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention; (5) QTc>480ms (QTc interval is calculated using the Fridericia formula; if QTc is abnormal, it can be detected continuously three times every 2 minutes, and the average value is taken).
9. History of spontaneous rupture of liver tumors.
10. Individuals with a history of hepatic encephalopathy.
11. Congenital or acquired immune dysfunction in subjects (such as HIV infected individuals).
12. There have been incidents of thrombosis or embolism occurring within the first 6 months of treatment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
13. Participants with a history of gastrointestinal bleeding or a clear tendency towards gastrointestinal bleeding within 6 months prior to the start of the study treatment, such as those at risk of bleeding or severe esophageal and gastric varices, locally active gastrointestinal ulcer lesions, or continuous positive fecal occult blood, cannot be included in the study. (If fecal occult blood is positive during the baseline period, a follow-up examination is required. If the follow-up examination is still positive, gastroduodenoscopy (EGD) is required. If EGD indicates a risk of bleeding, esophageal and gastric varices/other gastrointestinal diseases cannot be included in the study.)
14. Within 6 months prior to the start of treatment, there have been abdominal fistulas, gastrointestinal perforation, or abdominal abscesses.
15. Severe, unhealed or cracked wounds, as well as active ulcers or untreated fractures.
16. Known genetic or acquired bleeding (such as coagulation dysfunction) or thrombotic tendencies, such as in hemophilia participants; Currently or recently (within 10 days prior to the start of research treatment), full dose oral or injection anticoagulants or thrombolytic drugs (prophylactic use of low-dose aspirin, low molecular weight heparin allowed) have been used for therapeutic purposes.
17. Major vascular diseases (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) occur within 6 months prior to the surgery.
18. Severe infection within 4 weeks prior to the surgery, including but not limited to hospitalization due to complications of infection, bacteremia, or severe pneumonia; Oral or intravenous administration of therapeutic antibiotics within 2 weeks prior to the start of the study treatment (subjects who receive prophylactic antibiotics, such as preventing urinary tract infections or exacerbation of chronic obstructive pulmonary disease, are eligible to participate in the study).
19. Use immunosuppressive agents or systemic hormone therapy within 14 days prior to the surgery to achieve immunosuppressive effects (dose>10mg/day prednisone or other therapeutic hormones).
20. Received attenuated live vaccine treatment within 28 days prior to the surgery.
21. According to the judgment of the researchers, the subjects may have other factors that may affect the research results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious illnesses (including mental illness) that require concurrent treatment, serious laboratory test abnormalities, and family or social factors that may affect the safety of the subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with hepatocellular carcinoma who have received immunotherapy based neoadjuvant or conversion therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Perioperative risk | From enrollment to the end of surgery at 4 weeks
  The criteria for perioperative risk include four aspects: operation time, transfusion, postoperative hospital stay, and complication. Operation time >200min is counted as 3 points, transfusion is counted as 2 points, postoperative hospital stay >8 days is counted as 2 points, and complication is counted as 1 point. The total score range is 0-8 points. Participants with a score of 3 or lower are considered to have a low perioperative risk, while those above 3 are considered to have a high perioperative risk.

SECONDARY OUTCOMES:
Progression free survival time | From enrollment to the end of surgery at 12 months
  The time between the end of surgery and tumor progression ( in any way ) or death ( for any reason )
Overall survival time | From enrollment to the end of surgery at 36 months
  The time from the end of surgery to death ( for any reason )

CONTACTS AND LOCATIONS:
Overall Officials: Tao Li, Principal Investigator — Shandong University
Locations (1):
- Qilu hospital of Shandong university, Jinan, Shandong, China